CLINICAL TRIAL: NCT02250560
Title: An Open Study to Investigate the Safety and Efficacy of Replenine®-VF by Continuous Infusion in Haemophilia B Patients Undergoing Major Surgery.
Brief Title: A Study to Investigate the Safety and Efficacy of Replenine®-VF in Haemophilia B Patients Undergoing Major Surgery.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Other Study IDs: R9VFCIMS
Record Dates: First submitted 2014-09-02; First posted 2014-09-26 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2014-08

CONDITIONS: Haemophilia B
MeSH Terms: conditions — Hemophilia B

ARMS (1):
- Replenine®-VF (Experimental)
  Interventions: Biological: Replenine®-VF (High Purity Factor IX)

INTERVENTIONS:
Biological: Replenine®-VF (High Purity Factor IX)

SUMMARY:
The main objective of the study is to investigate the safety and efficacy of Replenine®-VF administered by continuous infusion in appropriate dosage to prevent bleeding and achieve haemostasis in patients with haemophilia B undergoing major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe Haemophilia B (≤5% baseline Factor IX level) due to undergo major surgery, previously treated patients, at least 16 years of age without inhibitors, currently receiving Factor IX concentrate.

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-04; Primary Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Assessment of control of prevention of bleeding | End of study (Day 5 to Day 10)
  Investigator's assessment as excellent, good, moderate or none.

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - North Hampshire Haemophilia Centre, Uplands House, North Hampshire Hospital, Aldermaston Road, Basingstoke
  - Haemophilia Centre, The Royal London Hospital, White Chapel, London
  - Haemophilia Centre and Haemostasis Unit, Royal Free Hospital, Pond Street, London
  - Manchester Thrombosis and Haemostasis Centre, University of Manchester, Department of Haematology, Manchester Royal Infirmary, Oxford Road, Manchester
  - Haemophilia Centre, Southampton General Hospital, Tremona Road, Southampton

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk